CLINICAL TRIAL: NCT05071872
Title: Retrospective Post-Market Clinical Follow Up of Rotarex®S & Aspirex®S Catheters in Treating Thrombotic Occlusion of Arteriovenous Graft for Dialysis Access (Artificial Bypass)
Brief Title: PMCF of Rotarex®S & Aspirex®S Catheters in Treating Thrombotic Occlusion of Arteriovenous Graft
Status: Completed | Type: Observational
Sponsor: Straub Medical AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-Arteriovenous Graft
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2021-12

CONDITIONS: Arteriovenous Graft Thrombosis
MeSH Terms: interventions — Atherectomy; Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rotarex®S: Treatment performed with Rotarex®S
  Interventions: Device: Atherectomy/Thrombectomy
- Aspirex®S: Treatment performed with Aspirex®S
  Interventions: Device: Atherectomy/Thrombectomy

INTERVENTIONS:
Device: Atherectomy/Thrombectomy — Percutaneous transluminal removal of thrombotic occlusion in arteriovenous graft

SUMMARY:
Retrospective Post-Market Clinical Follow Up of Rotarex®S & Aspirex®S Catheters in treating thrombotic occlusion of Arteriovenous Graft for dialysis access (Artificial Bypass)

DETAILED DESCRIPTION:
To evaluate the safety, technical performance, and clinical efficacy of the Rotarex®S & Aspirex®S Catheters as a stand-alone and adjunctive therapy for the treatment of acute thrombotic occlusion of arteriovenous graft for dialysis access (Artificial Bypass) in accordance with Rotarex®S & Aspirex®S Catheters intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subject with a minimum age of 18 years
2. Treatment performed between 2013 and 2020
3. Occlusion in arteriovenous graft
4. For the Rotarex®S group: use of Rotarex®S Catheter
5. For the Aspirex®S group: use of Aspirex®S Catheter

Exclusion Criteria:

1. Subjects not appropriate for this study according to the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute thrombotic occlusion of arteriovenous graft for dialysis access (Artificial Bypass) treated with either Rotarex®S Catheter nor Aspirex®S Catheter
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Technical success | Day 1
  defined as removal of thrombotic occlusion in AV-G with Rotarex®S or Aspirex®S Catheter

SECONDARY OUTCOMES:
Procedural success | Day 1
  defined as restoration of blood flow in AV-G following Rotarex®S or Aspirex®S Catheter ± adjunctive treatment
Successful use of AV-Graft as dialysis access | Up to 14 days
  Successful use of AV-Graft as dialysis access post-procedure on at least two occasions
Primary and Secondary Patency | 10 days, 1, 3 and 6 months
  defined as ability to perform dialysis at 10 days, 1 month, 3 months and 6 months
(SAEs) Serious Adverse events Rate | 6 months
  SAEs as defined per ISO 14155
Procedure-related Adverse events Rate | 6 months
  Procedure-related AEs as defined per ISO 14155
(ADEs) Adverse device effects Rate | 6 months
  Adverse device effects (ADEs) as defined per ISO 14155
(SADEs) Serious Adverse Device Effects Rate | 6 months
  (SADEs) Serious Adverse Device Effects as defined per ISO 14155

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Heller, M.D., Principal Investigator — Angiocentrum Příbram
Locations (1):
- Angiocentrum Příbram, Příbram, Czechia